CLINICAL TRIAL: NCT03668496
Title: A Phase III, Randomized,Double-Blind, Multi-center Study to Investigate the Efficacy and Safety of SHR-1210 in Combination With Carboplatin and Paclitaxel Versus Placebo in Combination With Carboplatin and Paclitaxel in First-Line Stage IV Squamous Non-Small Cell Lung Cancer
Brief Title: A Study of SHR-1210 in Combination With Carboplatin + Paclitaxel in Subjects With Squamous NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-307
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer Squamous Cell; Lung Cancer Stage IV; PD-1 Antibody; Chemotherapy Effect
MeSH Terms: conditions — Lung Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 +chemotherapy (Experimental): subject will receive SHR-1210 200mg every 3 weeks, carboplatin AUC 5 on Day 1 of each 21 day, 4-6 cycles Paclitaxel 175mg/m2, Day 1 of each 21 day, 4-6 cycles
  Interventions: Drug: SHR-1210
- chemotherapy (Active Comparator): carboplatin AUC 5 on Day 1 of each 21 day, 4-6 cycles Paclitaxel 175mg/m2, Day 1 of each 21 day, 4-6 cycles
  Interventions: Drug: The placebo

INTERVENTIONS:
Drug: SHR-1210 — Drug delivery cycle is 3 weeks, and in the experimental group,200 mg shr-1210 was given with Carboplatin and Paclitaxel in the first day of each cycle, with intravenous drip.
  Arms: SHR-1210 +chemotherapy
Drug: The placebo — in the control group,placebo was given with Carboplatin and Paclitaxel in the first day of each cycle, with intravenous drip.
  Arms: chemotherapy

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, multicenter phase III clinical study. Target population is patients with stage IV squamous non-small cell lung cancer who had not received systemic chemotherapy. Study objective is to compare the efficacy and safety of SHR-1210 + carboplatin + paclitaxel with placebo + carboplatin + paclitaxel in study population in China. SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subject will be randomized into study arm or control arm to accept study treatment. Subjects who randomized into control will have the opportunity to receive cross over treatment of SHR-1210 monotherapy after confirmed disease progression. Treatment cycles of chemotherapy will be 4-6 which will be decided by investigators.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with histopathological diagnosis of squamous non-small cell lung cancer (SqNSCLC) and clinical stage IV
2. has not received prior systemic treatment for metastatic NSCLC.
3. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status
4. Has archived Tumor tissue samples
5. Subject must have a measurable target lesion based on RECIST v1.1 .
6. Has adequate organ function.
7. Women of childbearing age must undergo a serological pregnancy test within 7 days before the first dose with negative results. Female subjects of reproductive age and male subjects whose spouse is a woman of reproductive age must agree to effective contraception within 180 days after the study period and the last dose of the study drug.
8. Subjects should be voluntarily participate in clinical studies and informed consent should be signed.

Exclusion Criteria:

1. active brain metastases and meningeal metastasis
2. uncontrollable tumor-related pain
3. massive pleural effusion, peritoneal effusion or pericardial effusion which cannot be controlled by repeated drainage;
4. radiotherapy to lung that is >30 Gy within 24 weeks before the first dose,
5. imaging (CT or MRI) showed that the tumor invading the large vessels
6. Known EGFR/ALK mutation.
7. subjects with any known or suspected autoimmune diseases
8. subjects with known or suspected interstitial pneumonia;
9. Subjects with severe cardiovascular and cerebrovascular diseases
10. arteriovenous thrombosis events, such as deep vein thrombosis and pulmonary embolism, occurred within 3 months;
11. female subjects who are pregnant or lactation or who plan to be pregnant during the study period;
12. positive HIV test;
13. active hepatitis B
14. evidence of active TB infection within 1 year before first dose;
15. severe infection occurred within 4 weeks before the first dose
16. patients with clinically significant bleeding symptoms or with obvious bleeding tendency in the first month
17. subjects who is on systemic immunogenic agents;
18. a history of severe allergic reactions to other monoclonal antibodies/fusion proteins;
19. History of severe allergic reactions to carboplatin or paclitaxel or their preventive drugs;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 month
  PFS, defined as the time from randomization to the first occurrence of disease progression as determined by the Independent Review Committee according to RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free survival | up to 24 month
  Progression-free survival (PFS) assessed by investigators according to RECIST V 1.1
Overall Survival (OS) | up to 24 month
  defined as time from the randomized to the time of the patient's death from any reason assessed by researchers.
Objective Response Rate (ORR) | up to 24 month
  The percentage of patients with CR and PR assessed by investigators according to Recist v 1.1.
disease control rate (DCR) | up to 24 month
  The proportion of patients who have achieved complete response， partial response and Stable disease assessed by investigators according to Recist v 1.1.
Duration of response （DoR） | up to 24 month
  According to Recist v 1.1 accessed by investigators
Adverse events (AEs) | up to 24 month
  All adverse event/Serious adverse event that occurred during the study period according to CTCAE v 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zou, MD, PhD, Study Director — Jiangsu HengRui Medicine Co., Ltd.; Caicun Zhou, MD, PhD, Principal Investigator — Tongji University, Shanghai Pulmonary Hospital
Locations (52):
- China (52):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA Ceneral Hospital, Beijing, Beijing Municipality
  - The Seventh Medical Center of PLA Ceneral Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - 900TH Hospital of Joint Logistics Support Force, Fuzhou, Fujian
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated Hospital of Chengde Medical College, Chengde, Hebei
  - The Fourth Hospital of Hebei Medical University (Hebei Cancer Hospital), Shijiazhuang, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Tongji Hospital, Tongji Medical College of Hust, Wuhan, Hubei
  - Xiang yang Central Hospital, Xiangyang, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital Of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Jinan Central Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Tongji University, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Shaanxi Provincial Cancer Hospital, Xian, Shanxi
  - Sichuan Provincial Cancer Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan
  - The First Affiliated Hospital，ZheJiang University, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital ZheJiang University School Of Medicine, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University of Medicine, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jiang T, Chen J, Xu X, Cheng Y, Chen G, Pan Y, Fang Y, Wang Q, Huang Y, Yao W, Wang R, Li X, Zhang W, Zhang Y, Hu S, Guo R, Shi J, Wang Z, Cao P, Wang D, Fang J, Luo H, Geng Y, Xing C, Lv D, Zhang Y, Yu J, Cang S, Zhang Y, Zhang J, Yang Z, Shi W, Zou J, Zhou C, Ren S. On-treatment blood TMB as predictors for camrelizumab plus chemotherapy in advanced lung squamous cell carcinoma: biomarker analysis of a phase III trial. Mol Cancer. 2022 Jan 3;21(1):4. doi: 10.1186/s12943-021-01479-4. PMID 34980131
- [Derived] Ren S, Chen J, Xu X, Jiang T, Cheng Y, Chen G, Pan Y, Fang Y, Wang Q, Huang Y, Yao W, Wang R, Li X, Zhang W, Zhang Y, Hu S, Guo R, Shi J, Wang Z, Cao P, Wang D, Fang J, Luo H, Geng Y, Xing C, Lv D, Zhang Y, Yu J, Cang S, Yang Z, Shi W, Zou J, Zhou C; CameL-sq Study Group. Camrelizumab Plus Carboplatin and Paclitaxel as First-Line Treatment for Advanced Squamous NSCLC (CameL-Sq): A Phase 3 Trial. J Thorac Oncol. 2022 Apr;17(4):544-557. doi: 10.1016/j.jtho.2021.11.018. Epub 2021 Dec 16. PMID 34923163